CLINICAL TRIAL: NCT00691288
Title: Effect of Omega-3 Fatty Acid Supplementation on Hypertriglyceridemia in HIV-infected Children Taking Highly Active Antiretroviral Therapy (HAART): a Randomized Cross-over Study
Brief Title: Effect of Omega-3 Fatty Acid Supplementation on Hypertriglyceridemia in HIV-infected Children
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to enroll sufficient patients
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Foundation for AIDS Research (CANFAR) (Other); The Physicians' Services Incorporated Foundation (Other); Ocean Nutrition (Industry)
Responsible Party: Principal Investigator, Ari Bitnun, Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1000011295
Record Dates: First submitted 2008-05-27; First posted 2008-06-05 (Estimated); Last update posted 2014-06-12 (Estimated); Status verified 2014-06

CONDITIONS: Hypertriglyceridemia
Keywords: omega-3 fatty acid; hypertriglyceridemia; HIV; pediatric; HAART
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Omega Pure followed by placebo
- 2 (Experimental)
  Interventions: Drug: Placebo followed by Omega Pure

INTERVENTIONS:
Drug: Omega Pure followed by placebo — Subjects in this arm will begin the study on active capsules (containing Omega Pure). Subjects in the 5-11 age group will take 2 capsules containing 500mg EPA/DHA twice daily for 12 weeks. Subjects in the 12-18 age group will take 2 capsules containing 1.0g EPA/DHA twice daily, also for a period of 12 weeks. Both age groups will then be switched to the placebo capsules containing citrus-flavoured soybean and corn oil, identical in appearance to the active agent, to be taken on an identical regimen to the active pills, for a period of 12 weeks.
  Other Names: omega-3 fatty acid supplementation
  Arms: 1
Drug: Placebo followed by Omega Pure — Patients assigned to this arm of the study will begin on placebo followed by Omega Pure (identical dose and regimen as arm 1), also for a period of 12 weeks each.
  Other Names: Omega-3 fatty acid supplementation
  Arms: 2

SUMMARY:
The overall objective of this study is to evaluate the safety and efficacy of fish oil omega-3-fatty acid supplementation in treating pediatric HAART-associated hypertriglyceridemia.

DETAILED DESCRIPTION:
There are no guidelines as to the clinical threshold at which treatment for hypertriglyceridemia is necessary in pediatric populations, and extreme hypertriglyceridemia is relatively infrequent in HIV-infected children. Adult studies have suggested that there is a proportionate reduction in triglycerides of approximately 15-25% when taking fish oil omega-3 fatty acid supplementation, irrespective of the degree of initial triglyceride elevation. This trial would thus represent a proof-of-concept study in children with mild to moderate hypertriglyceridemia.

The results of this study would contribute to the pool of knowledge regarding the efficacy and safety of this nutriceutical in the treatment of HAART-associated hypertriglyceridemia in children. Compared with other interventions (such as dietary changes and drug therapies), nutritional supplementation with fish oil is an inexpensive, simple, and likely preferable treatment for a potentially significant medical condition. In addition, the results of this study could presumably be extrapolated to benefit children with hypertriglyceridemia secondary to other types of drugs or illnesses.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive children aged 5-18 years on stable HAART therapy for at least 6 months, with reasonable control of their HIV (viral load remaining undetectable, or stable with <0.5 log increase in previous 3-4 months) and no plans for a change in therapy in the next year
* Elevated fasting triglyceride level >1.5 mmol/L on at least two occasions within the previous year (including at least one in the last 3 months while on the current HAART regimen)
* Ability to swallow capsules

Exclusion Criteria:

* Known allergy to fish, soybean, or corn
* Current treatment with triglyceride-lowering agent
* Family history of familial hypertriglyceridemia

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2008-06; Primary Completion 2011-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Percentage change in triglyceride levels | 4 and 12 weeks after beginning treatment

SECONDARY OUTCOMES:
Changes in cholesterol profiles (LDL, HDL, and total:HDL ratio), amylase, platelet function, AST, and ALT | 4 and 12 weeks after beginning treatment
Reporting of side effects, compliance, and discontinuation | 4 and 12 weeks after beginning treatment
Effect on control of HIV (vial load, CD4) | 12 weeks after beginning treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ari Bitnun, MD, MSc, Principal Investigator — The Hospital for Sick Children; Jason Brophy, MD, Principal Investigator — The Hospital for Sick Children; Stanley Read, MD, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada